CLINICAL TRIAL: NCT03716700
Title: Real-world CANadian CUvitru Non-Interventional Study in Subjects Transitioning From Subcutaneous Immunoglobulin (CANCUN)
Status: Completed | Type: Observational
Sponsor: Baxalta now part of Shire (Industry)
Collaborators: Baxalta Innovations GmbH, now part of Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Other Study IDs: SHP664-402
Record Dates: First submitted 2018-08-31; First posted 2018-10-23 (Actual); Last update posted 2021-03-05 (Actual); Status verified 2021-03

CONDITIONS: Primary Immunodeficiency Diseases (PID)
MeSH Terms: conditions — Primary Immunodeficiency Diseases | interventions — Hizentra; Solutions; gamma-Globulins

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Cohort 1: Cohort1 will include the participants who have been transitioned to CUVITRU at the time of enrollment in the study.
  Interventions: Biological: CUVITRU
- Cohort 2: Cohort 2 will include participants 6 months (±2 weeks) after CUVITRU initiation.
  Interventions: Biological: CUVITRU
- Cohort 3: Cohort 3 will include participants 12 months (-1 or +2 months) after CUVITRU initiation.
  Interventions: Biological: CUVITRU

INTERVENTIONS:
Biological: CUVITRU — CUVITRU
  Other Names: 20% Solution; IGSC; Immune Globulin Subcutaneous (Human)

SUMMARY:
This study will provide insights on the infusion parameters, dosing, and experience of participants transitioning to CUVITRU in a real-world setting.

ELIGIBILITY:
Inclusion Criteria (The participant will not be considered eligible for the study without meeting all of the criteria below):

* Voluntarily provide written, signed, and dated (personally or via a legally authorized representative) informed consent or assent as applicable to participate in the study;
* Participant > 2 years of age with a documented diagnosis of PID or SID requiring IgG replacement therapy, as defined by the International Union of Immunological Societies Scientific Committee 2009 and by diagnostic criteria according to Conley et al., 1999;
* Participant has received subcutaneous immunoglobulin (SCIG) therapy previous to CUVITRU for at least 3 months; and
* Participant has received CUVITRU in line with the product specification (CUVITRU Product Monograph (Baxalta Canada Corporation, 2018) at start of study

Exclusion Criteria (Participants are excluded from the study if any of the following criteria are met):

* Participation in any interventional clinical study within the last 30 days
* Participant participates in a clinical study in parallel during the observation period; and
* Participant had a dose change 30 days prior to transition to CUVITRU for Cohort 1

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Data will be collected on approximately 500 participants with primary immunodeficiency (PID) and secondary immunodeficiency (SID) requiring Immunoglobulin G (IgG) replacement therapy across 8-10 sites in Canada (excluding Quebec). Any specific number of participants in each cohort is not a requirement.
Sampling Method: Non-Probability Sample
Enrollment: 126 (Actual)
Dates: Start 2018-09-24 (Actual); Primary Completion 2020-07-23 (Actual); Study Completion 2020-07-23 (Actual)

PRIMARY OUTCOMES:
Infusion parameter 1: Cohort 1-Start of data collection | Baseline
  Median infusion volume per site
Infusion parameter 1: Cohort 1- Month 3 | Month 3
  Median infusion volume per site
Infusion parameter 1: Cohort 1- Month 6 | Month 6
  Median infusion volume per site
Infusion parameter 1: Cohort 1- 12 Month final follow-up | 12 Month final follow-up
  Median infusion volume per site
Infusion parameter 1: Cohort 2- Start of data collection | Baseline
  Median infusion volume per site
Infusion parameter 1: Cohort 2- 12 Month final follow-up | 12 Month final follow-up
  Median infusion volume per site
Infusion parameter 1.1: Cohort 1- Start of data collection | Baseline
  Median infusion volume per infusion
Infusion parameter 1.1: Cohort 1- Month 3 | Month 3
  Median infusion volume per infusion
Infusion parameter 1.1: Cohort 1- Month 6 | Month 6
  Median infusion volume per infusion
Infusion parameter 1.1: Cohort 1- 12 Month final follow-up | 12 Month final follow-up
  Median infusion volume per infusion
Infusion parameter 1.1: Cohort 2- Start of data collection | Baseline
  Median infusion volume per infusion
Infusion parameter 1.1: Cohort 2- 12 Month final follow-up | 12 Month final follow-up
  Median infusion volume per infusion
Infusion parameter 2: Cohort 1- Start of data collection | Baseline
  Median number of infusion sites
Infusion parameter 2: Cohort 1- Month 3 | Month 3
  Median number of infusion sites
Infusion parameter 2: Cohort 1- Month 6 | Month 6
  Median number of infusion sites
Infusion parameter 2: Cohort 1- 12 Month final follow-up | 12 Month final follow-up
  Median number of infusion sites
Infusion parameter 2: Cohort 2- Start of data collection | Baseline
  Median number of infusion sites
Infusion parameter 2: Cohort 2- 12 Month final follow-up | 12 Month final follow-up
  Median number of infusion sites
Infusion parameter 3: Cohort 1- Start of data collection | Baseline
  Median infusion duration
Infusion parameter 3: Cohort 1- Month 3 | Month 3
  Median infusion duration
Infusion parameter 3: Cohort 1- Month 6 | Month 6
  Median infusion duration
Infusion parameter 3: Cohort 1- 12 Month final follow-up | 12 Month final follow-up
  Median infusion duration
Infusion parameter 3: Cohort 2- Start of data collection | Baseline
  Median infusion duration
Infusion parameter 3: Cohort 2- 12 Month final follow-up | 12 Month final follow-up
  Median infusion duration
Infusion parameter 3.1: Cohort 1- Month 3 Follow-up | Month 3
  Median number of infusions to reach participant's maximum infusion volume
Infusion parameter 3.1: Cohort 1- Month 6 Follow-up | Month 6
  Median number of infusions to reach participant's maximum infusion volume
Infusion parameter 3.1: Cohort 1- 12 Month final follow-up | 12 Month final follow-up
  Median number of infusions to reach participant's maximum infusion volume
Infusion parameter 3.1: Cohort 2- 12 Month final follow-up | 12 Month final follow-up
  Median number of infusions to reach participant's maximum infusion volume
Infusion parameter 3.2: Cohort 1- Start of data collection | Baseline
  Median number of infusions per month per participant
Infusion parameter 3.2: Cohort 1- Month 3 | Month 3
  Median number of infusions per month per participant
Infusion parameter 3.2: Cohort 1- Month 6 | Month 6
  Median number of infusions per month per participant
Infusion parameter 3.2: Cohort 1- 12 Month final follow-up | 12 Month final follow-up
  Median number of infusions per month per participant
Infusion parameter 3.2: Cohort 2- Start of data collection | Baseline
  Median number of infusions per month per participant
Infusion parameter 3.2: Cohort 2- 12 Month final follow-up | 12 Month final follow-up
  Median number of infusions per month per participant
Infusion parameter 3.3: Cohort 1- Start of data collection | Baseline
  Median number of infusions to reach final dose interval per participant
Infusion parameter 3.3: Cohort 1- Month 3 | Month 3
  Median number of infusions to reach final dose interval per participant
Infusion parameter 3.3: Cohort 1- Month 6 | Month 6
  Median number of infusions to reach final dose interval per participant
Infusion parameter 3.3: Cohort 1- 12 Month final follow-up | 12 Month final follow-up
  Median number of infusions to reach final dose interval per participant
Infusion parameter 3.3: Cohort 2- Start of data collection | Baseline
  Median number of infusions to reach final dose interval per participant
Infusion parameter 3.3: Cohort 2- 12 Month final follow-up | 12 Month final follow-up
  Median number of infusions to reach final dose interval per participant
Infusion parameter 1: Cohort 3- 12 Month Final Follow-up | 12 Month final follow-up
  Median infusion volume per site.
Infusion parameter 1.1: Cohort 3- 12 Month Final Follow-up | 12 Month final follow-up
  Median infusion volume per infusion.
Infusion parameter 2: Cohort 3- 12 Month final follow-up | 12 Month final follow-up
  Median number of infusion sites.
Infusion parameter 3: Cohort 3- 12 Month final follow-up | 12 Month final follow-up
  Median infusion duration.
Infusion parameter 3.1: Cohort 3- 12 Month final follow-up | 12 Month final follow-up
  Median number of infusions to reach participant's maximum infusion volume (infusion rate)
Infusion parameter 3.2: Cohort 3- 12 Month final follow-up | 12 Month final follow-up
  Median number of infusions per month per participant
Infusion parameter 3.3: Cohort 3- 12 Month final follow-up | 12 Month final follow-up
  Median number of infusions to reach final dose interval per participant

SECONDARY OUTCOMES:
Infusion parameter 4.1: Cohort 1- Start of data collection | Baseline
  Median maximal infusion rate per site
Infusion parameter 4.1: Cohort 1- Month 3 | Month 3
  Median maximal infusion rate per site
Infusion parameter 4.1: Cohort 1- Month 6 | Month 6
  Median maximal infusion rate per site
Infusion parameter 4.1: Cohort 1- 12 Month final follow-up | 12 Month final follow-up
  Median maximal infusion rate per site
Infusion parameter 4.1: Cohort 2- Start of data collection | Baseline
  Median maximal infusion rate per site
Infusion parameter 4.1: Cohort 2- 12 Month final follow-up | 12 Month final follow-up
  Median maximal infusion rate per site
Infusion parameter 4.2: Cohort 1- Start of data collection | Baseline
  Number of infusions that are discontinued, slowed, or interrupted
Infusion parameter 4.2: Cohort 1- Month 3 | Month 3
  Number of infusions that are discontinued, slowed, or interrupted
Infusion parameter 4.2: Cohort 1- Month 6 | Month 6
  Number of infusions that are discontinued, slowed, or interrupted
Infusion parameter 4.2: Cohort 1- 12 Month final follow-up | 12 Month final follow-up
  Number of infusions that are discontinued, slowed, or interrupted
Infusion parameter 4.2: Cohort 2- Start of data collection | Baseline
  Number of infusions that are discontinued, slowed, or interrupted
Infusion parameter 4.2: Cohort 2- 12 Month final follow-up | 12 Month final follow-up
  Number of infusions that are discontinued, slowed, or interrupted
Infusion parameter 4.3: Cohort 1- Month 3 | Month 3
  Median number of infusions to reach participant's maximum infusion rate
Infusion parameter 4.3: Cohort 1- Month 6 | Month 6
  Median number of infusions to reach participant's maximum infusion rate
Infusion parameter 4.3: Cohort 1- 12 Month final follow-up | 12 Month final follow-up
  Median number of infusions to reach participant's maximum infusion rate
Infusion parameter 4.3: Cohort 2- 12 Month final follow-up | 12 Month final follow-up
  Median number of infusions to reach participant's maximum infusion rate
Infusion parameter 5.1: Cohort 1- Start of data collection | Baseline
  Mean dose
Infusion parameter 5.1: Cohort 1- Month 3 | Month 3
  Mean dose
Infusion parameter 5.1: Cohort 1- Month 6 | Month 6
  Mean dose
Infusion parameter 5.1: Cohort 1- 12 Month final follow-up | 12 Month final follow-up
  Mean dose
Infusion parameter 5.1: Cohort 2- Start of data collection | Baseline
  Mean dose
Infusion parameter 5.1: Cohort 2- 12 Month final follow-up | 12 Month final follow-up
  Mean dose
Infusion parameter 5.2: Cohort 1- Start of data collection | Baseline
  Mean dosing interval
Infusion parameter 5.2: Cohort 1- Month 3 | Month 3
  Mean dosing interval
Infusion parameter 5.2: Cohort 1- Month 6 | Month 6
  Mean dosing interval
Infusion parameter 5.2: Cohort 1- 12 Month final follow-up | 12 Month final follow-up
  Mean dosing interval
Infusion parameter 5.2: Cohort 2- Start of data collection | Baseline
  Mean dosing interval
Infusion parameter 5.2: Cohort 2- 12 Month final follow-up | 12 Month final follow-up
  Mean dosing interval
Infusion parameter 5.3: Cohort 1- Start of data collection | Baseline
  Mean number of dose adjustments
Infusion parameter 5.3: Cohort 1- Month 3 | Month 3
  Mean number of dose adjustments
Infusion parameter 5.3: Cohort 1- Month 6 | Month 6
  Mean number of dose adjustments
Infusion parameter 5.3: Cohort 1- 12 Month final follow-up | 12 Month final follow-up
  Mean number of dose adjustments
Infusion parameter 5.3: Cohort 2- Start of data collection | Baseline
  Mean number of dose adjustments
Infusion parameter 5.3: Cohort 2- 12 Month final follow-up | 12 Month final follow-up
  Mean number of dose adjustments
Infusion parameter 4.1: Cohort 3- 12 Month final follow-up | 12 Month final follow-up
  Median maximal infusion rate per site
Infusion parameter 4.2: Cohort 3- 12 Month final follow-up | 12 Month final follow-up
  Number of infusions that are discontinued, slowed, or interrupted
Infusion parameter 4.3: Cohort 3- 12 Month final follow-up | 12 Month final follow-up
  Median number of infusions to reach participant's maximum infusion rate
Infusion parameter 5.1: Cohort 3- 12 Month final follow-up | 12 Month final follow-up
  Mean dose
Infusion parameter 5.2: Cohort 3- 12 Month final follow-up | 12 Month final follow-up
  Mean dosing interval
Infusion parameter 5.3: Cohort 3- 12 Month final follow-up | 12 Month final follow-up
  Mean number of dose adjustments
Treatment Satisfaction Questionnaire for Medication-9 (TSQM-9): Cohort 1 | 12 Month final follow-up
  TSQM-9 is a 9-item, validated, self-administered instrument used to assess participant's satisfaction with medication. The three domains assessed are effectiveness (3 items), convenience (3 items), and global satisfaction (3 items). Scores for each domain are calculated by adding up the items in each domain and then transforming the composite score into a value ranging from 0 to 100. Higher score indicated greater satisfaction in that domain.
Treatment Satisfaction Questionnaire for Medication-9 (TSQM-9): Cohort 2 | 12 Month final follow-up
  TSQM-9 is a 9-item, validated, self-administered instrument used to assess participant's satisfaction with medication. The three domains assessed are effectiveness (3 items), convenience (3 items), and global satisfaction (3 items). Scores for each domain are calculated by adding up the items in each domain and then transforming the composite score into a value ranging from 0 to 100. Higher score indicated greater satisfaction in that domain.
Treatment Satisfaction Questionnaire for Medication-9 (TSQM-9): Cohort 3 | 12 Month final follow-up
  TSQM-9 is a 9-item, validated, self-administered instrument used to assess participant's satisfaction with medication. The three domains assessed are effectiveness (3 items), convenience (3 items), and global satisfaction (3 items). Scores for each domain are calculated by adding up the items in each domain and then transforming the composite score into a value ranging from 0 to 100. Higher score indicated greater satisfaction in that domain.
Life Quality Index (LQI): Cohort 1 | 12 Month final follow-up
  The LQI is a self-administered questionnaire developed specifically for participants/legal guardians involved in IVIG treatments. It consists of 15-items, divided into four domains: treatment interferences (6 items), therapy-related problems (4 items), therapy setting (3 items), and treatment costs (2 items). Items are rated on a 7-point Likert-type scale ranging from 1: "Extremely bad" to 7: "Extremely good". Total scores range from 15 to 105, with higher scores indicating the highest possible satisfaction with factors such as independence, therapy convenience, social/school/work activities, and health and travel costs.
Life Quality Index (LQI): Cohort 2 | 12 Month final follow-up
  The LQI is a self-administered questionnaire developed specifically for participants/legal guardians involved in IVIG treatments. It consists of 15-items, divided into four domains: treatment interferences (6 items), therapy-related problems (4 items), therapy setting (3 items), and treatment costs (2 items). Items are rated on a 7-point Likert-type scale ranging from 1: "Extremely bad" to 7: "Extremely good". Total scores range from 15 to 105, with higher scores indicating the highest possible satisfaction with factors such as independence, therapy convenience, social/school/work activities, and health and travel costs
Life Quality Index (LQI): Cohort 3 | 12 Month final follow-up
  The LQI is a self-administered questionnaire developed specifically for participants/legal guardians involved in IVIG treatments. It consists of 15-items, divided into four domains: treatment interferences (6 items), therapy-related problems (4 items), therapy setting (3 items), and treatment costs (2 items). Items are rated on a 7-point Likert-type scale ranging from 1: "Extremely bad" to 7: "Extremely good". Total scores range from 15 to 105, with higher scores indicating the highest possible satisfaction with factors such as independence, therapy convenience, social/school/work activities, and health and travel costs
Treatment Preference Questionnaire (TPQ): Cohort 1 | 12 Month final follow-up
  The TPQ is a self-administered questionnaire developed to assess participants' preference towards the administration of new subcutaneous immunoglobulin G (SCIG) therapy.
  There are 4-items on the questionnaire, which investigate a participant's reference on the clinic/hospital/home setting of receiving the immunoglobulin therapy, the participant's rating on the frequency and method of administration, and the participant's preference to continue receiving the SCIG treatment.
Treatment Preference Questionnaire (TPQ): Cohort 2 | 12 Month final follow-up
  The TPQ is a self-administered questionnaire developed to assess participants' preference towards the administration of new subcutaneous immunoglobulin G (SCIG) therapy. There are 4-items on the questionnaire, which investigate a participant's preference on the clinic/hospital/home setting of receiving the immunoglobulin therapy, the participant's rating on the frequency and method of administration, and the participant's preference to continue receiving the SCIG treatment.
Treatment Preference Questionnaire (TPQ): Cohort 3 | 12 Month final follow-up
  The TPQ is a self-administered questionnaire developed to assess participants' preference towards the administration of new subcutaneous immunoglobulin G (SCIG) therapy. There are 4-items on the questionnaire, which investigate a participant's preference on the clinic/hospital/home setting of receiving the immunoglobulin therapy, the participant's rating on the frequency and method of administration, and the participant's preference to continue receiving the SCIG treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Shire
Locations (3):
- Canada (3):
  - University of McMaster, Hamilton, Ontario
  - Grand River Allergy, Kitchener, Ontario
  - Toronto Allergists, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- [Derived] Keith PK, Cowan J, Kanani A, Kim H, Lacuesta G, Lee JK, Chen J, Park M, Gladiator A. Transitioning subcutaneous immunoglobulin 20% therapies in patients with primary and secondary immunodeficiencies: Canadian real-world study. Allergy Asthma Clin Immunol. 2022 Aug 7;18(1):70. doi: 10.1186/s13223-022-00709-8. PMID 35934726
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/5f6b5fe84db2bf003ab47afc